CLINICAL TRIAL: NCT05213390
Title: A Clinical Investigation of an Autonomous Phone Conversational Agent for Cataract Surgery Follow-up
Brief Title: Autonomous Telephone Follow-up After Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Collaborators: University of Oxford (Other); Imperial College London (Other)
Responsible Party: Principal Investigator, Edward Meinert, PhD, Evaluation Lead, University of Plymouth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21WE6780
Record Dates: First submitted 2021-11-08; First posted 2022-01-28 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Cataract; After Cataract
MeSH Terms: conditions — Cataract; Capsule Opacification

STUDY DESIGN:
Intervention Model Description: The study will be a multi-centre, mixed-methods clinical investigation to develop evidence regarding the feasibility, acceptability and potential effectiveness of Dora.
Masking Description: No masking is possible, because all participants receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dora follow-up phone call (Experimental): DORA uses a variety of AI technologies to deliver the patient follow-up call, including: speech transcription, natural language understanding, a machine-learning conversation model to enable contextual conversations, and speech generation. Together, these technologies cover the input, processing and analysis, and output needed to maintain a natural conversation. DORA is configured to deliver calls through a telephone connection as a real-time, stand-alone system: the operator inputs individual patient details to initiate the call and completes a summary in the electronic health record (EHR) afterwards. The entire conversation will be supervised by a clinician. This clinician will be able to interrupt the call at any point if the system fails, the patient struggles to interact with it, or DORA does not collect sufficient information from the patient. The clinician will record a clinical assessment which will be compared to the DORA assessment.
  Interventions: Other: Dora

INTERVENTIONS:
Other: Dora — DORA uses a variety of AI technologies to deliver the patient follow-up call, including: speech transcription, natural language understanding, a machine-learning conversation model to enable contextual conversations, and speech generation. Together, these technologies cover the input, processing and analysis, and output needed to maintain a natural conversation. DORA is configured to deliver calls through a telephone connection as a real-time, stand-alone system: the operator inputs individual patient details to initiate the call and completes a summary in the electronic health record (EHR) afterwards.

SUMMARY:
This project will apply AI technology to meet the gap between increasing demand and limited capacity of high- volume healthcare services. The project will develop evidence that will support the safe deployment of Ufonia's automated telemedicine platform to deliver calls to cataract surgery patients at two large NHS hospital trusts.

The proposed study will implement DORA in addition to the current standard of care for a cohort of patients at Imperial College Healthcare Trust and Oxford University Hospitals NHS Foundation Trust. The study will evaluate the agreement of DORA's decision with an expert clinician. In addition it will test the acceptability of the solution for patients and clinicians; the sensitivity and specificity of the system in deciding if a patient requires additional review; and the health economic benefits of the solution to patients (reduced time and travel) and the local healthcare system. If successful, a proposal will be developed to roll the solution out to all patients at each site in anticipation of an application to a late phase award for wider NHS deployment.

DETAILED DESCRIPTION:
Background

Due to an ageing population and increased expectation, the demand for many services is exceeding the capacity of the clinical workforce. As a result, staff are facing a crisis of burnout from being pressured to deliver high- volume workloads, driving increasing costs for providers. Artificial intelligence, in the form of conversational agents, presents a possible opportunity to enable efficiencies in the delivery of care.

Aims and Objectives

This study aims to evaluate the effectiveness, usability and acceptability of DORA - an AI-enabled autonomous telemedicine call - for detection of post-operative cataract surgery patients who require further assessment. The study's objectives are: to establish efficacy of DORA's decision making in comparison to an expert human clinician; baseline sensitivity and specificity for detection of true complications; evaluation of patient acceptability; evidence for cost-effectiveness; and to capture data that may support further studies.

Project plan and methods used

Based on implementation science, the interdisciplinary study will be a mixed-methods phase one pilot establishing inter-observer reliability; as well as usability and acceptability.

Timelines for delivery

The study will last eighteen months: seven months of evaluation and intervention refinement, nine months of implementation and follow-up, and two months of post-evaluation analysis and write-up.

Anticipated Impact and Dissemination

The project's key contributions will be evidence on artificial intelligence voice conversational agent effectiveness, and associated usability and acceptability. Results will be disseminated in peer-reviewed journals and at international medical sciences and engineering conferences.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent;
* Aged 18 years or older;
* On the waiting list for routine cataract surgery. Cataract surgery as part of a combined procedure with other ocular surgery will not be included;
* No history or presence of significant ocular comorbidities that would be expected to alter the risks of cataract surgery or normal post-operative follow-up schedule. Note that significant ocular comorbidities do not include stable, chronic, or inactive ocular conditions such as amblyopia, drop-controlled stable glaucoma or ocular hypertension, previous squint surgery, inactive macular pathology, previous refractive surgery, or previous vitreoretinal surgery with stable retina.

Exclusion Criteria:

* Individuals with any condition that could preclude the ability to comply with the study or follow-up procedures;
* Presence of ocular or systemic uncontrolled disease (unless deemed not clinically significant by the Investigator and Sponsor);
* Involved in current research related to this technology or been involved in related research to this technology prior to recruitment;
* Cognitive difficulties, hearing impairment or non-English speakers;
* History of current or severe, unstable or uncontrolled systemic disease (unless deemed not clinically significant by the Investigator and Sponsor).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Normando, MD, PhD, Study Chair — Imperial College London
Locations (2):
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

REFERENCES:
- [Background] Milne-Ives M, de Cock C, Lim E, Shehadeh MH, de Pennington N, Mole G, Normando E, Meinert E. The Effectiveness of Artificial Intelligence Conversational Agents in Health Care: Systematic Review. J Med Internet Res. 2020 Oct 22;22(10):e20346. doi: 10.2196/20346. PMID 33090118
- [Background] de Pennington N, Mole G, Lim E, Milne-Ives M, Normando E, Xue K, Meinert E. Safety and Acceptability of a Natural Language Artificial Intelligence Assistant to Deliver Clinical Follow-up to Cataract Surgery Patients: Proposal. JMIR Res Protoc. 2021 Jul 28;10(7):e27227. doi: 10.2196/27227. PMID 34319248
- [Derived] Milne-Ives M, Homer SR, Andrade J, Meinert E. Mapping the Process of Engagement With Digital Health Interventions: A Cross-Case Synthesis. Mayo Clin Proc Innov Qual Outcomes. 2025 May 27;9(3):100625. doi: 10.1016/j.mayocpiqo.2025.100625. eCollection 2025 Jun. PMID 40503087
- [Derived] Meinert E, Milne-Ives M, Lim E, Higham A, Boege S, de Pennington N, Bajre M, Mole G, Normando E, Xue K. Accuracy and safety of an autonomous artificial intelligence clinical assistant conducting telemedicine follow-up assessment for cataract surgery. EClinicalMedicine. 2024 Jul 3;73:102692. doi: 10.1016/j.eclinm.2024.102692. eCollection 2024 Jul. PMID 39050586

RESULTS

PARTICIPANT FLOW:
Groups:
- Dora Follow-up Phone Call: DORA uses a variety of AI technologies to deliver the patient follow-up call, including: speech transcription, natural language understanding, a machine-learning conversation model to enable contextual conversations, and speech generation. DORA is configured to deliver calls through a telephone connection as a real-time, stand-alone system: the operator inputs individual patient details to initiate the call and completes a summary in the electronic health record (EHR) afterwards. The entire conversation will be supervised by a clinician. This clinician will be able to interrupt the call at any point if the system fails, the patient struggles to interact with it, or DORA does not collect sufficient information from the patient. The clinician will record a clinical assessment which will be compared to the DORA assessment.
  Dora: DORA uses a variety of AI technologies to deliver the patient follow-up call, including: speech transcription, natural language understanding, a machine-learning conversation model to enable contextual conversations, and speech generation. Together, these technologies cover the input, processing and analysis, and output needed to maintain a natural conversation. DORA is configured to deliver calls through a telephone connection as a real-time, stand-alone system: the operator inputs individual patient details to initiate the call and completes a summary in the electronic health record (EHR) afterwards.
Period: Overall Study
Arm/Group | Dora Follow-up Phone Call
Started | 225
Completed | 202
Not Completed | 23
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 12
Not completed — Protocol Violation | 9

BASELINE CHARACTERISTICS:
Arm/Group | Dora Follow-up Phone Call
Number analyzed (Participants) | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Ethnicity data was not available for 2 participants.
  Participants
    Ethnicity: number analyzed (Participants) | 200
    Ethnicity: White | 160
    Ethnicity: Asian | 12
    Ethnicity: Black | 11
    Ethnicity: Other | 17
First or second cataract surgery [Count of Participants; unit: Participants]
  First eye | 113
  Second eye | 89
Income [Count of Participants; unit: Participants] — Population: Not all participants completed the self-report questionnaire or provided data for every item
  Participants
    number analyzed (Participants) | 147
    ≤ £19,999/yr | 28
    £20,000-29,999/yr | 24
    £30,000-39,999/yr | 5
    £40,000-49,999/yr | 5
    £50,000-69,999/yr | 9
    >£70,000/yr | 6
    Undefined | 70
Education level [Count of Participants; unit: Participants] — Population: Not all participants completed the self-report questionnaire or provided data for every item
  Participants
    number analyzed (Participants) | 131
    Lower Than Bachelor's Degree | 88
    Bachelor's Degree or Higher | 43

OUTCOME MEASURES:

1. Primary Outcome: Agreement
Description: Inter-rater reliability: the degree of agreement between DORA and the clinician on their assessments of the individual symptoms and the management plan; Whether or not the clinician had to interrupt the call to ask clarifying questions
Time Frame: Inter-rater reliability was assessed based on data collected during Dora calls, which lasted an average of 7.5 minutes
Population: Calls to 7 of the 202 were incomplete.
Measure: Count of Participants; unit: Participants
Groups:
- Dora Outcome Decision: Dora's decision about whether the participant could be discharged after their call without requiring further clinician assessment.
- Supervising Clinician Decision: The supervising clincian's decision about whether the participant could be discharged after their call without requiring further clinician assessment.
Arm/Group | Dora Outcome Decision | Supervising Clinician Decision
Number analyzed (Participants) | 195 | 195
Participants
  Discharge | 117 | 131
  Review | 78 | 64

2. Secondary Outcome: Clinical Complications Identified or Missed by DORA System
Description: Clinical data was collected from patients' electronic health record (EHR) up to 90 days postoperatively to capture numbers of participants 'recommended discharge' by Dora R1 with subsequent unexpected management change
Time Frame: Up to 90 days post surgery
Measure: Count of Participants; unit: Participants
Groups:
- Unexpected Management Change: Of the patients for whom Dora's decision recommended discharge after their call without requiring further clinician assessment, how many had a subsequent unexpected management change that occurred within 90 days of the surgery.
Arm/Group | Unexpected Management Change
Number analyzed (Participants) | 117
Participants | 10

3. Secondary Outcome: Calls Completed Without Intervention
Description: Number of autonomous calls that were completed without needing any intervention from the supervising clinician; Clinician-reported reasons for asking clarifying questions
Time Frame: Dora calls lasted an average of 7.5 minutes
Measure: Number; unit: DORA follow-up calls
Arm/Group | Dora Follow-up Phone Call
Number analyzed (Participants) | 202
DORA follow-up calls
  Call completed autonomously | 195
  Call incomplete | 7

4. Secondary Outcome: System Usability
Description: Measured using the System Usability Scale (minimum of 0, maximum of 100, higher scores indicate better usability)
Time Frame: Usability assessments were completed up to 6 months after the Dora call
Population: Not all participants completed the usability questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dora Follow-up Phone Call
Number analyzed (Participants) | 131
units on a scale | 77.76 (17.55)

5. Secondary Outcome: Usability of Telehealth System Implementation
Description: Measured using the Telehealth Usability Questionnaire (minimum score of 1, maximum score of 5, averaged across 19 items; higher scores indicate better usability)
Time Frame: Usability was assessed up to 6 months after the call
Population: Not all participants completed the usability questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dora Follow-up Phone Call
Number analyzed (Participants) | 115
units on a scale | 3.79 (0.89)

6. Secondary Outcome: Qualitative Patient Perspectives of Usability
Description: Qualitative feedback from semi-structured interviews
Time Frame: Semi-structured interview call, lasting up to 30 minutes, conducted up to 6 months after the Dora call
Population: Participants invited for semi-structured interviews - categories reflect major components of the Theoretical Framework of Acceptability and the number of participants who provided feedback that was coded into those categories.
Measure: Number; unit: participants
Groups:
- Dora Follow-up Phone Call: DORA uses a variety of AI technologies to deliver the patient follow-up call, including: speech transcription, natural language understanding, a machine-learning conversation model to enable contextual conversations, and speech generation. Together, these technologies cover the input, processing and analysis, and output needed to maintain a natural conversation. DORA is configured to deliver calls through a telephone connection as a real-time, stand-alone system: the operator inputs individual patient details to initiate the call and completes a summary in the electronic health record (EHR) afterwards.
Arm/Group | Dora Follow-up Phone Call
Number analyzed (Participants) | 20
participants
  Burden | 18
  Opportunity costs | 12
  Self-efficacy | 5
  Intervention coherence | 17

7. Secondary Outcome: Acceptability of AI Follow-up Phone Call
Description: Qualitative feedback from semi-structured interviews
Time Frame: Semi-structured interview call, lasting up to 30 minutes, conducted up to 6 months after the Dora call
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Dora Follow-up Phone Call
Number analyzed (Participants) | 20
participants
  Affective attitude (anticipated) | 15
  Affective attitude (experienced) | 20
  Ethicality | 5

8. Secondary Outcome: Satisfaction With AI Follow-up Phone Call
Description: Qualitative feedback from semi-structured interviews
Time Frame: Semi-structured interview call, lasting up to 30 minutes, conducted up to 6 months after the Dora call
Population: Interviewed participants were asked if they would be willing to use Dora again; their responses were coded into the three categories below.
Measure: Number; unit: participants
Arm/Group | Dora Follow-up Phone Call
Number analyzed (Participants) | 20
participants
  Willing | 15
  Not willing | 1
  Hesitant, but willing | 4

9. Secondary Outcome: Appropriateness of AI for Follow-up Assessment
Description: Qualitative feedback from semi-structured interviews
Time Frame: Semi-structured interview call, lasting up to 30 minutes, conducted up to 6 months after the Dora call
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Dora Follow-up Phone Call
Number analyzed (Participants) | 20
participants
  Perceived effectiveness (anticipated) | 4
  Perceived effectiveness (experienced) | 19
  Perceived effectiveness (long-term) | 19

10. Secondary Outcome: Cost Impact
Description: A cost analysis compared the direct costs of face-to-face (F2F) follow-up at Imperial with Dora R1 (in Oxford, patients do not have routine postoperative follow-up). Assumptions included annual costs for various healthcare professionals and the duration of F2F follow-up appointments (estimated at 30 min).
Time Frame: Conducted 6 months after baseline
Population: Patients on the Imperial post-cataract surgery pathway
Measure: Number; unit: Great British Pounds
Arm/Group | Dora Follow-up Phone Call
Number analyzed (Participants) | 97
Great British Pounds
  Total staff cost (standard pathway) | 4555.16
  Total staff cost (Dora pathway): number analyzed (Participants) | 92
  Total staff cost (Dora pathway) | 1084.21

11. Secondary Outcome: Subsequent Unplanned Follow-up
Description: Clinical data was collected from patients' electronic health record (EHR) up to 90 days postoperatively to capture numbers of participants 'recommended discharge' by Dora R1 with subsequent unplanned review.
Time Frame: Up to 90 days post surgery
Measure: Count of Participants; unit: Participants
Groups:
- Unplanned Follow-up: Of the patients for whom Dora's decision recommended discharge after their call without requiring further clinician assessment, how many had a subsequent unplanned follow-up that occurred within 90 days of the surgery.
Arm/Group | Unplanned Follow-up
Number analyzed (Participants) | 117
Participants | 5

ADVERSE EVENTS:
Time Frame: Up to 3 months post cataract surgery
Arm/Group | Dora Follow-up Phone Call
All-Cause Mortality (participants affected / at risk) | 0/202
Serious Adverse Events (participants affected / at risk) | 0/202
Other Adverse Events (participants affected / at risk) | 4/202
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dora Follow-up Phone Call (N=202)
Symptomatic patients with unexpected management changes (Eye disorders) | 4 — For patients who 'passed' their phone assessment, but were found to be symptomatic at follow-up with unexpected management changes apart from lubricants or advice, such as surgical intervention and additional specialist follow-up or investigations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT05213390/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT05213390/SAP_001.pdf